CLINICAL TRIAL: NCT03315624
Title: Safety and Clinical Performance of a Dialyzer With a Modified Polysulfone Membrane - eMPORA Study (Modified POlysulfone membRAne)
Brief Title: Safety and Clinical Performance of a Dialyzer With a Modified Polysulfone Membrane
Acronym: eMPORA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HD-FX-05-EU
Record Dates: First submitted 2017-10-10; First posted 2017-10-20 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Renal Failure; End Stage Renal Disease
Keywords: Hemodialysis; Hemodiafiltration; Renal replacement therapy
MeSH Terms: conditions — Renal Insufficiency; Kidney Failure, Chronic | interventions — Kidneys, Artificial

STUDY DESIGN:
Intervention Model Description: Prospective, open, controlled, cross-over (with randomized treatment sequences), interventional, multi-center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemodiafiltration HDF (Other): Three consecutive treatment weeks and one follow-up week per patient. Each treatment week includes three hemodiafiltration sessions with the dialyzer FX CORAL 600 (TD 16-1), the dialyzer FX CorDiax 600 or the dialyzer FX 600. In each week the patient is assigned to one type of dialyzer.
  Interventions: Device: Dialyzer

INTERVENTIONS:
Device: Dialyzer — Three hemodiafiltration sessions assigned to one type of dialyzer FX Coral 600, FX 600 and FX CorDiax 600

SUMMARY:
The clinical investigation will be performed to generate clinical data on clearances and removal rates (for ß2-microglobulin, myoglobin, phosphate, creatinine, and urea) as well as biocompatibility of the modified polysulfone membrane to obtain CE-certification according to the European Medical Device Directive for the FX Coral 600 (TD 16-1) dialyzer.

DETAILED DESCRIPTION:
The FX Coral (TD 16-1) dialyzer is a new development with a modified polysulfone membrane and is not CE marked yet. The purpose of the clinical evaluation is to generate clinical data for the CE approval.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years
* Informed consent signed and dated by study patient and investigator / authorized physician
* Ability to understand the nature and requirements of the study

Exclusion Criteria:

* Any condition which could interfere with the patient's ability to comply with the study. This decision is at the discretion of the treating physician and relates to the general good condition of the patient (e.g. absence of any acute condition, e.g. infection or mental problem which might give reason for concern etc.).
* Ongoing participation in an interventional clinical study during the preceding 30 days
* Previous participation in this study
* Pregnancy (pregnancy test will be conducted with female patients aged less or aged 55 years) or lactation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2017-12-09 (Actual); Study Completion 2018-03-14 (Actual)

PRIMARY OUTCOMES:
Removal rate of 2-microglobulin | t=240 min. of HDF
  Removal rate of 2-microglobulin will be calculated as primary endpoint in blood samples to evaluate the clinical performance of the new FX Coral 600 (TD 16-1) dialyzer.

SECONDARY OUTCOMES:
Clearance of ß2-microglobulin | t=60 min. of HDF
Removal rates of myoglobin | t=240 min. of HDF
Clearances of myoglobin | t= 60 min. of HDF

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Wagner, Dr, Principal Investigator — Georg-Haas-Dialysezentrum der PHV, Giessen, Germany
Locations (1):
- Georg-Haas-Dialysezentrum der PHV, Giessen, Germany